CLINICAL TRIAL: NCT03692013
Title: Effect of Nighttime Losartan on Prognosis of Nocturnal Hypertension Patients Undergoing Continous Ambulatory Peritoneal Dialysis
Brief Title: Nighttime Losartan in Continous Ambulatory Peritoneal Dialysis (NVCAPD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cheng Wang, Director of Nephrology, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Losartan
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Hypertension,Nephropathy
Keywords: Nocturnal hypertension,Peritoneal dialysis,Losartan
MeSH Terms: conditions — Hypertensive Nephropathy | interventions — Losartan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nighttime group (Experimental): patients with nocturnal hypertension taking losartan at nighttime
  Interventions: Drug: Losartan
- daytime group (Active Comparator): patients with nocturnal hypertension taking losartan at daytime
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Participants will be divided into 2 groups as daytime group and nighttime group The participants in daytime group will take 100-200mg Losartan in the morning between 6AM to 8AM. The participants in nighttime group will take 100-200mg Losartan at night between 9PM to 11PM .
  Other Names: Cozaar

SUMMARY:
Hypertension is one of the most important independent risk factors for the prognosis of continous ambulatory peritoneal dialysis patients. The incident rate is high and the control rate is low. Nocturnal hypertension has been paid more attention in recent years. Compared to daytime blood pressure, nocturnal blood pressure is an independent and efficient prognostic indicator of hypertensive deaths and cardiovascular events, but it is lack of evidence about its impact on prognosis in peritoneal dialysis patients and the effective treatment program. Our previous cohort study suggests that the incidence of nocturnal hypertension in patients with chronic kidney disease is up to 71.22%, with a significant increase as the decline of renal function, and more severe target organ damage in patients with nocturnal hypertension: the decrease of glomerular filtration rate, left ventricular hypertrophy, and the increase of all cause death and cardiovascular death. Our small sample size study show that night time antihypertensive drugs can better control blood pressure and delay the development of left ventricular hypertrophy. These preliminary results suggest that nocturnal hypertension is closely related to the prognosis of chronic renal disease. Taking antihypertensive drugs at night is one of the options for controlling nocturnal hypertension. However, it is not clear whether taking antihypertensive drugs at night can improve the prognosis of maintenance peritoneal dialysis patients with nocturnal hypertension. To this end, the investigators collect continous ambulatory peritoneal dialysis patients with nocturnal hypertension, and propose a time selective use of losartan to intervene in nocturnal hypertension. By comparing the difference in the effects of losartan on the prognosis of maintenance peritoneal dialysis patients during the day or night, to further clarify the role of nocturnal hypertension in the prognosis of maintenance peritoneal dialysis patients, whether controlling nocturnal hypertension can improve the prognosis of maintenance peritoneal dialysis patients. The completion of study will optimize the prevention and treatment of hypertension in maintenance peritoneal dialysis patients, and provide an evidence for precise prevention and treatment of nocturnal hypertension in maintenance peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old and <75 years.
2. Diagnosed as chronic kidney disease 5th stage in accordance with the KDIGO guide 2012 (egfr < 15 ml/ (min 1.73m2)).
3. Accept 3-5 bags daily, continous ambulatory peritoneal dialysis for >3 months.
4. Ambulatory blood pressure monitoring indicates nighttime systolic blood pressure (SBP) > 120mmHg and / or diastolic blood pressure (DBP) > 70mmHg.

Exclusion Criteria:

1. Night learning or work, irregular rest for a long time.
2. Moderate and severe edema in difficult to correct
3. Persistent atrial fibrillation.
4. Severe anemia and severe dystrophy.
5. Patients with postural hypotension or symptomatic hypotension.
6. Severe side effects or contraindications of valsartan treatment.
7. Treatment of corticosteroids or other hormones at present.
8. Unable to cooperate or unable to tolerate ambulatory blood pressure monitoring.
9. Ineffective ambulatory blood pressure data.
10. The clinical data were incomplete during the treatment period; end-point events occurred within 6 months or follow-up time was less than 6 months.
11. In the first 3 months before admission, there were obvious cardiovascular and cerebrovascular diseases such as coronary syndrome, myocardial infarction or stroke.
12. There were complications such as vascular disease, infection and bleeding within 1 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 5 years
  Rate of death caused by all causes

SECONDARY OUTCOMES:
cardiovascular mortality | 5 years
  Rate of death caused by cardiovascular events, such as myocardial infarction,arrythmia and heart failure
cerebrovascular mortality | 5 years
  Rate of death caused by cerebral vascular events, such as stroke
incidence of cardiocerebral vascular events | 5 years
  Incidence of cardiovascular and cerebrovascular events that require hospitalization and lead to death or non death, including myocardial infarction, heart failure, stroke,vascular reconstruction,peripheral vascular disease, and non-traumatic amputation

OTHER OUTCOMES:
incidence of cardiovascular structural abnormalities | 5 years
  Incidence changes of carotid artery intima-media thickness and left ventricular mass index

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Wang, Director, Principal Investigator — Nephrology Department, the Fifth Affiliated Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jager KJ, Merkus MP, Dekker FW, Boeschoten EW, Tijssen JG, Stevens P, Bos WJ, Krediet RT. Mortality and technique failure in patients starting chronic peritoneal dialysis: results of The Netherlands Cooperative Study on the Adequacy of Dialysis. NECOSAD Study Group. Kidney Int. 1999 Apr;55(4):1476-85. doi: 10.1046/j.1523-1755.1999.00353.x. PMID 10201013
- [Background] Udayaraj UP, Steenkamp R, Caskey FJ, Rogers C, Nitsch D, Ansell D, Tomson CR. Blood pressure and mortality risk on peritoneal dialysis. Am J Kidney Dis. 2009 Jan;53(1):70-8. doi: 10.1053/j.ajkd.2008.08.030. Epub 2008 Nov 22. PMID 19027213
- [Background] Foley RN, Parfrey PS. Cardiovascular disease and mortality in ESRD. J Nephrol. 1998 Sep-Oct;11(5):239-45. PMID 9831236
- [Background] Cocchi R, Degli Esposti E, Fabbri A, Lucatello A, Sturani A, Quarello F, Boero R, Bruno M, Dadone C, Favazza A, Scanziani R, Tommasi A, Giangrande A. Prevalence of hypertension in patients on peritoneal dialysis: results of an Italian multicentre study. Nephrol Dial Transplant. 1999 Jun;14(6):1536-40. doi: 10.1093/ndt/14.6.1536. PMID 10383021
- [Background] Menon MK, Naimark DM, Bargman JM, Vas SI, Oreopoulos DG. Long-term blood pressure control in a cohort of peritoneal dialysis patients and its association with residual renal function. Nephrol Dial Transplant. 2001 Nov;16(11):2207-13. doi: 10.1093/ndt/16.11.2207. PMID 11682669
- [Background] Buckalew VM Jr, Berg RL, Wang SR, Porush JG, Rauch S, Schulman G. Prevalence of hypertension in 1,795 subjects with chronic renal disease: the modification of diet in renal disease study baseline cohort. Modification of Diet in Renal Disease Study Group. Am J Kidney Dis. 1996 Dec;28(6):811-21. doi: 10.1016/s0272-6386(96)90380-7. PMID 8957032
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force for the Management of Arterial Hypertension of the European Society of Hypertension and the European Society of Cardiology. 2013 ESH/ESC Practice Guidelines for the Management of Arterial Hypertension. Blood Press. 2014 Feb;23(1):3-16. doi: 10.3109/08037051.2014.868629. Epub 2013 Dec 20. No abstract available. PMID 24359485
- [Background] Hodgkinson J, Mant J, Martin U, Guo B, Hobbs FD, Deeks JJ, Heneghan C, Roberts N, McManus RJ. Relative effectiveness of clinic and home blood pressure monitoring compared with ambulatory blood pressure monitoring in diagnosis of hypertension: systematic review. BMJ. 2011 Jun 24;342:d3621. doi: 10.1136/bmj.d3621. PMID 21705406
- [Background] Parati G, Ochoa JE, Salvi P, Lombardi C, Bilo G. Prognostic value of blood pressure variability and average blood pressure levels in patients with hypertension and diabetes. Diabetes Care. 2013 Aug;36 Suppl 2(Suppl 2):S312-24. doi: 10.2337/dcS13-2043. No abstract available. PMID 23882065
- [Background] Mancia G, Zanchetti A, Agabiti-Rosei E, Benemio G, De Cesaris R, Fogari R, Pessina A, Porcellati C, Rappelli A, Salvetti A, Trimarco B. Ambulatory blood pressure is superior to clinic blood pressure in predicting treatment-induced regression of left ventricular hypertrophy. SAMPLE Study Group. Study on Ambulatory Monitoring of Blood Pressure and Lisinopril Evaluation. Circulation. 1997 Mar 18;95(6):1464-70. doi: 10.1161/01.cir.95.6.1464. PMID 9118514
- [Background] Cuspidi C, Sala C, Valerio C, Negri F, Mancia G. Nocturnal blood pressure in untreated essential hypertensives. Blood Press. 2011 Dec;20(6):335-41. doi: 10.3109/08037051.2011.587280. Epub 2011 Jun 9. PMID 21651423
- [Background] Hoshide S, Ishikawa J, Eguchi K, Ojima T, Shimada K, Kario K. Masked nocturnal hypertension and target organ damage in hypertensives with well-controlled self-measured home blood pressure. Hypertens Res. 2007 Feb;30(2):143-9. doi: 10.1291/hypres.30.143. PMID 17460384
- [Background] Yano Y, Kario K. Nocturnal blood pressure and cardiovascular disease: a review of recent advances. Hypertens Res. 2012 Jul;35(7):695-701. doi: 10.1038/hr.2012.26. Epub 2012 Mar 1. PMID 22378470
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Hansen TW, Li Y, Boggia J, Thijs L, Richart T, Staessen JA. Predictive role of the nighttime blood pressure. Hypertension. 2011 Jan;57(1):3-10. doi: 10.1161/HYPERTENSIONAHA.109.133900. Epub 2010 Nov 15. PMID 21079049
- [Background] Ortega LM, Materson BJ. Hypertension in peritoneal dialysis patients: epidemiology, pathogenesis, and treatment. J Am Soc Hypertens. 2011 May-Jun;5(3):128-36. doi: 10.1016/j.jash.2011.02.004. Epub 2011 Apr 1. PMID 21459067
- [Background] Kishi T, Hirooka Y, Konno S, Sunagawa K. Angiotensin II receptor blockers improve endothelial dysfunction associated with sympathetic hyperactivity in metabolic syndrome. J Hypertens. 2012 Aug;30(8):1646-55. doi: 10.1097/HJH.0b013e328355860e. PMID 22728908
- [Background] Pedro AA, Gehr TW, Brophy DF, Sica DA. The pharmacokinetics and pharmacodynamics of losartan in continuous ambulatory peritoneal dialysis. J Clin Pharmacol. 2000 Apr;40(4):389-95. doi: 10.1177/00912700022009099. PMID 10761166
- [Background] Wang C, Zhang J, Liu X, Li CC, Ye ZC, Peng H, Chen Z, Lou T. Effect of valsartan with bedtime dosing on chronic kidney disease patients with nondipping blood pressure pattern. J Clin Hypertens (Greenwich). 2013 Jan;15(1):48-54. doi: 10.1111/jch.12021. Epub 2012 Oct 9. PMID 23282124